CLINICAL TRIAL: NCT00448188
Title: Thrombocytes and International Normalized Ratio Are no Predictors for Bleeding in Application of Central Veneous Catheters
Brief Title: Bleeding Risk in CVCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bleeding risk in CVCs
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2007-09

CONDITIONS: Bleeding
Keywords: central venous catheter; international normalized ratio; thrombocytes; bleeding risk; all patients in need of central venous line; comparison of patients with normal hemostasis to such with disorders in hemostasis
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: central venous catheter application

SUMMARY:
Since many of the patients in an intensive care unit suffer from disorders of hemostasis, bleeding is a main concern applying central venous catheters. Even if there are some data indicating elevated international normalized ratio may not increase the risk of bleeding no clear cut-off has been defined so far. An INR > 1.5 is generally considered to increase the risk of bleeding. Furthermore, many authors consider platelets below 50 x 109 /l as a contra-indication to CVC cannulation, since there are some data this may increase the risk of bleeding. Therefore platelet transfusion before venous puncture is suggested. In our clinical experience INR > 1.5 and platelets < 50 x 109 /l do not correlate with increased risk of bleeding. The aim of this study is to demonstrate, that coagulopathy, defined by INR and platelet count, is not decisive for bleeding.

ELIGIBILITY:
Inclusion Criteria:

* All patients acquiring a central venous catheter

Exclusion Criteria:

* Patients pre or post surgery
* Patients with bleeding due to other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bleeding within 24 hours after cvc application
other complications within the first 24 hours

SECONDARY OUTCOMES:
mortality
long-term complications

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Weigand, Dr., Principal Investigator — University Hospital Heidelberg, Department of Gastroenterology, Heidelberg, Germany; Jens Encke, Prof. Dr., Study Director — University Hospital Heidelberg, Department of Gastroenterology, Heidelberg, Germany
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Weigand K, Encke J, Meyer FJ, Hinkel UP, Munder M, Stremmel W, Zahn A. Low levels of prothrombin time (INR) and platelets do not increase the risk of significant bleeding when placing central venous catheters. Med Klin (Munich). 2009 May 15;104(5):331-5. doi: 10.1007/s00063-009-1070-2. Epub 2009 May 16. PMID 19444412